CLINICAL TRIAL: NCT06533644
Title: A Phase 2a Multicenter, Dose-Escalation and Dose Optimization Study of SYNC-T Therapy SV-102 for Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: A Study of SYNC-T Therapy SV-102 in Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Syncromune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: LEGION-100-2a
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Intervention Model Description: Part 1 of the study is a dose escalation design followed by Part 2 randomized, blinded, dose optimization design.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1 - Dose Escalation, Cohort 1: Partial Oncolysis + SV-102 (Experimental): Participants will receive partial oncolysis plus an intratumoral infusion of SV-102, Dose Level 1.
  Interventions: Procedure: Partial Oncolysis; Drug: SV-102
- Part 1 - Dose Escalation, Cohort 2: Partial Oncolysis + SV-102 (Experimental): Participants will receive partial oncolysis plus an intratumoral infusion of SV-102, Dose Level 2.
  Interventions: Procedure: Partial Oncolysis; Drug: SV-102
- Part 1 - Dose Escalation, Cohort 3: Partial Oncolysis + SV-102 (Experimental): Participants will receive partial oncolysis plus an intratumoral infusion of SV-102, Dose Level 3.
  Interventions: Procedure: Partial Oncolysis; Drug: SV-102
- Part 2 - Dose Optimization, Arm 1: Partial Oncolysis + SV-102 (Experimental): Participants will receive partial oncolysis plus an intratumoral infusion of SV-102, dose level selected from Part 1.
  Interventions: Procedure: Partial Oncolysis; Drug: SV-102
- Part 2 - Dose Optimization, Arm 2: Partial Oncolysis + SV-102 (Experimental): Participants will receive partial oncolysis plus an intratumoral infusion of SV-102, dose level selected from Part 1.
  Interventions: Procedure: Partial Oncolysis; Drug: SV-102

INTERVENTIONS:
Procedure: Partial Oncolysis — Partial tumor oncolysis will be completed by cryolysis.
  Other Names: cryolysis
Drug: SV-102 — Intratumoral infusion of SV-102

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, and efficacy of SYNC-T Therapy SV-102 and to identify the maximum tolerated dose (MTD) and/or selected dose for phase 2b study.

ELIGIBILITY:
Inclusion Criteria:

* Male >=18 years old.
* Able to provide written informed consent and comply with the study procedures.
* Participants with advanced and/or metastatic histologically or cytologically confirmed adenocarcinoma of the prostate without small cell histology.
* Serum testosterone levels less than or equal to (<=) 0.5 nanograms per millilitre (ng/mL) (<=1.73 nanomoles per litre [nmol/L]) at screening if on anti-hormonal therapy.
* Progression after the receipt of one or more approved second-generation androgen-receptor-pathway inhibitors with or without a prior course of taxane therapy, and those who have not responded or progressed after standard therapies or for whom no further standard therapy exists or standard therapy is not available, and has not received more than three prior lines of therapy. If a poly adenosine diphosphate ribose (ADP)-ribose polymerase (PARP)-positive participants chose not to receive an approved PARP-inhibitor they will be eligible for the study.
* Able to undergo general anesthesia or conscious sedation.
* Has undergone a cardiac work-up and received cardiac clearance within 2 months before first treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of less than (<) 3.
* Life expectancy >=6 months
* Last dose of previous anticancer therapy (excluding hormonal therapy) must by 28 days or more prior to first study treatment.
* Resolution of all acute toxic effects (excluding alopecia) of any prior anticancer therapy.
* For males with female partners of childbearing potential, even if surgically sterilized (that is [i.e.], status post vasectomy), who agree to practice:

  1. effective barrier contraception during the treatment period and through 120-150 days after last dose, OR
  2. true abstinence, when this is in line with the preferred and usual lifestyle of the participants. Periodic abstinence (for example [e.g.], calendar, ovulation, symptothermal, post ovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.
* Has at least one lesion of at least 1 centimeter (cm), measurable in at least two dimensions within the prostate accessible transperineally using transrectal ultrasound (TRUS) that is demonstrable on magnetic resonance imaging (MRI)/computed tomography (CT) and is accessible for infusion on TRUS or, if a radical prostatectomy has been performed, has a metastatic lesion of at least 1 cm or lymph node lesion of at least 1.5 cm, that is demonstrable on MRI/CT and accessible by a percutaneous needle to permit both tumor biopsy and immunotherapy infusion. The eligible tumor lesion for intratumoral-infusion cannot be a tumor that is adjacent to vital structures such as major nerves or blood vessels or at risk of airway compromise in the event of post-infusion tumor swelling/inflammation.
* Participants receiving bone resorptive therapy must be on stable doses for at least 42 days prior to the oncolysis.
* In the opinion of the Investigator, there is no other meaningful life prolonging therapy option available, or the participant refuses other therapy, outside of anti-hormonal therapy.
* Adequate bone marrow, renal, and hepatic function.
* Participants agrees to provide tumor tissue and undergo an on-treatment tumor biopsy.

Exclusion Criteria:

* Has a known other primary malignancy other than prostate cancer that is progressing or has required active treatment in the last 3 years, excluding basal and squamous cell carcinoma, papillary thyroid cancer, and ductal carcinoma in situ of the breast.
* Has an obstructed urinary system before or after stenting.
* Has undergone major surgery, including local prostate intervention (excluding prostate biopsy), within 28 days prior to the first dose of study treatment and has not recovered adequately from the toxicities and/or complications.
* Has used any anticoagulants or other blood thinners pre-study treatments within the protocol-defined timelines.
* Has an active infection (including tuberculosis) requiring systemic therapy.
* Has a history of non-infectious pneumonitis that requires steroids.
* Has received a live vaccine within 30 days prior to the enrollment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 28 days prior to the first study treatment.
* Significant cardiac or other medical illness such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia (e.g., New York Heart Association Class 4), or history of previous heart failure.
* Fridericia corrected QT interval (QTcF) greater than (>) 470 millisecond (msec) (men) on a 12-lead electrocardiogram (ECG) during the screening period.
* Malignant pleural effusions or ascites that require immediate intervention.
* Brain metastases (includes history of).
* Prior history of autoimmune disease except hypothyroidism, uncontrolled or unmanaged diabetes (glycated haemoglobin [HbA1c] >=6.5), cardiac arrhythmia (unstable or untreated), hypersensitivity, or other illness or disease that in the opinion of the Principal Investigator, with consultation with Syncromune's Chief Medical Officer, makes the participant a poor candidate.
* History of bone marrow/stem cell transplant.
* Participants having human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS) are not eligible for enrollment.
* Active coronavirus disease-2019 (COVID-19) infection or tests positive for COVID-19 a day before or the day of planned study treatment.
* Participants who have active viral (any etiology) hepatitis are excluded.
* Participants with serologic evidence of chronic hepatitis B virus (HBV) infection (defined by a positive hepatitis B surface antigen [HBsAg] test and a positive hepatitis B core antibody (anti-HBc) test) who have a viral load below the limit quantification (HBV deoxyribonucleic acid [DNA] titer <1000 copies per milliliters [cps/mL] or 200 international units per milliliter [IU/mL]) and are not currently on viral suppressive therapy may be eligible and should be discussed with the Sponsor's Medical Monitor.
* Participants with a history of hepatitis C virus (HCV) infection should have completed curative antiviral treatment and have a viral load below the limit of quantification are eligible for study entry. Known or suspected hepatitis C infection which has not been treated and cured are not eligible. Known or suspected hepatitis C currently on treatment with an undetectable viral load are eligible. Patients with a history of hepatitis C virus (HCV) infection should have completed curative antiviral treatment and have a viral load below the limit of quantification are eligible for study entry.
* Participants with complications or contraindications related to the liver, including intrahepatic biliary ductal dilation, uncorrectable bleeding diathesis, and decompensated liver failure, tumor burden of over 5 lesions, tumors greater than 5 cm in size, tumors in close proximity to vital structures, such as portal vein, biliary tree, or gastrointestinal tract.
* Breast cancer gene (BRCA) mutation testing will be required for participants not previously treated with a PARP inhibitor, unless BRCA status is established prior to screening. If PARP-positive and participants agree to PARP therapy, they will be ineligible.
* Any condition(s) that, in the opinion of the Investigator, would increase the risk for toxicities from study treatment, or interfere with participants compliance or conduct of this study.
* Known visceral metastases.
* Known substance abuse or medical, psychological, or social conditions that may interfere with patient's participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-12-14 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Immune-related Adverse Reactions (imARs) | Up to 2 years
Maximum Tolerated Dose | Up to 48 weeks
  The MTD will be defined as the highest dose level below the dose level at which 2 or more participant experience a dose limiting toxicity (DLT).
Optimal Biologic Dose (OBD) | Up to 48 weeks
  OBD will be determined based on DLT and dose escalation part data.
Recommended Phase 2 Dose (RP2D) | Up to 48 weeks
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for the expansion phase, based on data collected during the dose escalation portion of the study.
Objective Response Rate (ORR) | Up to 2 years
  The ORR is defined as the percentage of participants who achieved best overall response (BOR) of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Duration of Response | Up to 2 years
  The period from the onset of a response (e.g., tumor shrinkage or stabilization) until disease progression or death, whichever occurs first.
Radiographic Progression-Free Survival (rPFS) per RECIST v1.1 and Prostate Cancer Working Group 3 (PCWG3) | Up to 2 years
  rPFS is defined as the time from the start of study drug until first documented radiologic disease progression at the first site of disease or death from any cause, whichever comes first.
Progression-Free Survival (PFS) | Up to 2 years
  The time interval between the start of treatment and the occurrence of disease progression or death from any cause.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from the first dose of study drug to death due to any cause.
Trough Concentration (Ctrough) of SV-102 | Pre-infusion at Day 1 of Cycle 1 up to Cycle 12 (each cycle length = 28 days)
Area Under the Concentration Time Curve From Time 0 to the Time t (AUC0-t) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Area Under the Concentration Time Curve From Time 0 to the Last Measurable Concentration (AUC0-last) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Maximum Observed Plasma Concentration (Cmax) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Last Observed (Quantifiable) Concentration (Clast) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Time to Reach the Maximum Plasma Concentration (Tmax) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Time of Last Measurable Concentration (Tlast) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Apparent Terminal Elimination Half-life (T1/2) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Apparent Total Body Clearance (CL/F) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Volume of Distribution (Vd) of SV-102 | Cycle 1: Pre-infusion up to 672 hours post-infusion; Cycle 3: Pre-infusion up to 72 hours post-infusion (each cycle length = 28 days)
Number of Participants With Any Device Constituent Failures/Malfunctions | Up to 2 years
Number of Participants With Anti-drug Antibodies (ADA) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Link, MD, Study Director — Syncromune, Inc.
Locations (5):
- United States (5):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Michigan Institute of Urology, Troy, Michigan
  - Mercy Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No